CLINICAL TRIAL: NCT03484104
Title: Cerebral Perfusion During Cardiac Surgery With Hypothermic Circulatory Arrest
Brief Title: Cerebral Perfusion in Hypothermic Circulatory Arrest
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Gabor Erdös, Consultant, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 2017-02216
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cerebrovascular Circulation
Keywords: Cardiopulmonary bypass; Hypothermic circulatory arrest; Aortic arch surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypothermic circulatory arrest: Patients undergoing cardiac surgery with hypothermic circulatory arrest and selective antegrade cerebral perfusion
  Interventions: Diagnostic Test: Measurement of tissue oxygenation index (TOI)

INTERVENTIONS:
Diagnostic Test: Measurement of tissue oxygenation index (TOI) — TOI and Vmca measurement during cardiac surgery with hypothermic circulatory arrest
  Other Names: Measurement of mean blood flow velocity in the middle cerebral artery (Vmca)

SUMMARY:
Selective antegrade cerebral perfusion (sACP) during aortic arch surgery in hypothermic circulatory arrest (HCA) is an established method for intraoperative neuroprotection. Although sACP is established as a beneficial method to reduce secondary neurological side effects due to brain-malperfusion, there are several parameters like sACP flow rate, perfusion pressure or temperature of the perfusate, where the optimal values remain unclear. The flow rate of the sACP-perfusate is increased according to center-specific standard-procedures. The optimal sACP flow rate, monitored by near infrared spectroscopy (NIRS), is to be investigated in this single center clinical prospective observational study. 40 Patients are enrolled over an estimated period of 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Elective cardiac surgery with cardiopulmonary bypass
* Hypothermic circulatory arrest
* General informed consent signed

Exclusion Criteria:

- Severe stenotis in cerebral arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population scheduled for elective aortic arch surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
TOI | through study completion, an average of 1 year
  The primary outcome is the tissue oxygenation index (TOI: NIRS value) at sACP flow rates of 6 , 8 and 10 (ml/kg/min) in comparison to the TOI measured awake.

SECONDARY OUTCOMES:
Vmca | through study completion, an average of 1 year
  The secondary outcome is the mean blood flow velocity in the middle cerebral artery at sACP the specified flow rates in comparison to the VmMCA during general anesthesia, after anesthesia induction.
Neurologic accidents | through study completion, an average of 1 year
  An additional secondary outcome measure are any neurologic accidents during the same hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD PhD, Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - Inselspital, University Hospital Bern, University of Bern, Bern
  - University of Bern, Bern

IPD SHARING:
Plan to Share IPD: No